CLINICAL TRIAL: NCT07168473
Title: A Randomized, Double-blind, Active-controlled, Parallel, Multi-center, Phase 3 Trial to Compare and Evaluate the Efficacy and Safety of DW1807 and DW1807-R2 in Perennial Allergic Rhinitis Patients With Asthma
Brief Title: Study to Evaluate the Efficacy and Safety of DW1807 in Perennial Allergic Rhinitis Patients With Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1807-301
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Perennial Allergic Rhinitis Accompanied by Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): DW1807 & DW1807-R2 placebo
  Interventions: Drug: Experimental
- Comparator (Active Comparator): DW1807 placebo & DW1807-R2
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Experimental — 1. DW1807 Once daily with water regardless of meals without chewing or crushing for up to 4 weeks
  2. DW1807-R2 placebo Once daily with water regardless of meals without chewing or crushing for up to 4 weeks
  Arms: Experimental
Drug: Comparator — 1. DW1807 placebo Once daily with water regardless of meals without chewing or crushing for up to 4 weeks
  2. DW1807-R2 Once daily with water regardless of meals without chewing or crushing for up to 4 weeks
  Arms: Comparator

SUMMARY:
This study aims to compare the efficacy and safety of DW1807 and DW1807-R2 in patients with perennial allergic rhinitis and comorbid asthma. The primary objective is to demonstrate the superiority of DW1807 over DW1807-R2 in improving the reflective total nasal symptom score (rTNSS) after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

<Screening Visit>

1. Male or female adults aged 19 years or older.
2. Individuals with a confirmed history or treatment record of perennial allergic rhinitis for at least 2 years at the time of screening.
3. Individuals who have a positive result on an allergy skin prick test or serum allergen-specific IgE antibody test (e.g., MAST or ImmunoCAP) conducted within 1 year prior to screening, and have a documented history of allergy to at least one perennial allergen (e.g., house dust mites, cats, dogs, molds, etc.).
4. Individuals diagnosed with asthma classified as Step 2 to Step 4.
5. Individuals who voluntarily provide written informed consent to participate in this clinical trial.

<Randomization Visit>

1. Subjects who meet all of the following criteria based on self-assessed nasal symptom scores recorded in the subject diary during the 7-day run-in period.

   ① Performed nasal symptom evaluations twice daily (morning and evening) on at least 4 days during the run-in period.

   ② Had an average daily Reflective Total Nasal Symptom Score (rTNSS) of ≥6 (maximum score: 12).
2. Subjects with medication compliance of ≥80% during the 7-day run-in period.

Exclusion Criteria:

<A. Disease and Medical History-Related Exclusion Criteria>

1. Individuals diagnosed with non-allergic rhinitis of other causes.
2. Individuals with a documented acute exacerbation of asthma within 12 weeks prior to screening.
3. Individuals diagnosed with pulmonary diseases other than asthma.
4. Individuals diagnosed with the following types of sinusitis:

   ① Acute sinusitis within 4 weeks prior to screening.

   ② Clinically significant chronic sinusitis, as determined by the investigator.
5. Individuals with nasal polyps or other clinically significant nasal structural abnormalities.
6. Individuals who have undergone nasal or perinasal surgery within 12 weeks prior to screening.
7. Individuals with a documented upper respiratory tract infection (including the common cold) or systemic infection within 3 weeks prior to screening.

<B. Concomitant Medication Use>

1. Subjects who have initiated immunotherapy or changed the dosage within 4 weeks prior to the screening visit.
2. Subjects who are on chronic use of medications that, in the opinion of the investigator, may interfere with the assessment of the investigational product's efficacy (e.g., tricyclic antidepressants).
3. Subjects who are currently taking, or are expected to require during the study, any medications that are prohibited as per the protocol.

<C. Laboratory Criteria>

1. Subjects with serum AST (GOT) or ALT (GPT) levels > 2 × the upper limit of normal (ULN) based on screening test results.
2. Subjects with an estimated glomerular filtration rate (eGFR, calculated by CKD-EPI) < 30 mL/min/1.73 m² based on screening test results.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
The mean change in reflective Total Nasal Symptom Score (rTNSS) | During the last 2 weeks of the treatment period (i.e., Weeks 3 to 4 of investigational product administration

SECONDARY OUTCOMES:
The mean change from baseline in reflective Total Nasal Symptom Score (rTNSS) | During the first two weeks of the treatment period (Weeks 1 through 2 of investigational product administration).
The mean change from baseline in instantaneous Total Nasal Symptom Score (iTNSS) | During both the first two weeks (Weeks 1 through 2) and the final two weeks (Weeks 3 through 4) of the treatment period.
The mean change from baseline in Daytime Nasal Symptom Score (DNSS) | During both the first two weeks (Weeks 1 through 2) and the final two weeks (Weeks 3 through 4) of the treatment period.
The mean change from baseline in Nighttime Nasal Symptom Score (NNSS) | During both the first two weeks (Weeks 1 through 2) and the final two weeks (Weeks 3 through 4) of the treatment period.
The mean change from baseline in Nighttime Symptom Score (NSS) | During both the first two weeks (Weeks 1 through 2) and the final two weeks (Weeks 3 through 4) of the treatment period.
The mean change from baseline in [Insert Specific Symptom or Score] | During both the first two weeks (Weeks 1 through 2) and the final two weeks (Weeks 3 through 4) of the treatment period.
The Global Evaluation of Allergic Rhinitis (GEAR) assessed independently by both the investigator and the subject | At Week 4 of investigational product administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No